# Artificiell intelligens - för att förutse och undvika blodtrycksfall under kirurgi

# Information till forskningspersoner

Vi vill fråga dig om du vill delta i ett forskningsprojekt. I det här dokumentet får du information om projektet och om vad det innebär att delta.

# Vad är det för ett projekt och varför vill ni att jag ska delta?

Det finns ett påvisat samband mellan blodtrycksfall i samband med operation och risken för att drabbas av komplikationer efteråt. Tyvärr är dessa episoder av blodtrycksfall svåra att förutse med de standardövervakningsmetoder som finns tillgängliga.

**Syftet med studien** är att med hjälp av artificiell intelligens (AI) bygga upp ett varningssystem som känner av när blodtrycket är på väg att sjunka redan innan blodtrycksfallet har inträffat. Ett sådant system skulle varna i god tid så att förebyggande behandling kan ges vilket skulle kunna minska risken för blodtrycksfall och påföljande komplikationer efter operation.

Ansökan är godkänd av Etikprövningsmyndigheten, diarienummer för prövningen hos Etikprövningsmyndigheten är 2022–06063

## Hur går projektet till?

Om du samtycker till att delta kommer du att opereras som planerat och övervakas enligt vår rutin. Vi kommer att samla in dina blodtrycksvärden, EKG, syresättning och övriga data som ingår i den standardövervakning vi använder under och efter operationen. Dessa data kommer vi sedan att använda för att bygga upp en AI-algoritm som kan förutspå blodtrycksfall.

#### Skillnader

Du sövs med en annan narkosmetod som innebär att du får sömnmedel och smärtstillande intravenöst (direkt i blodet) under operationen, istället för den standardmetod som vi använder vid operation i buken, dvs att narkos-gas tillsätts i inandningsluften. Intravenös narkos och smärtstillning är en väl beprövad metod som används vid flera andra typer av kirurgi.

I stället för en vanlig narkosapparat kommer en speciellt anpassad respirator användas för att stötta din andning. Denna respirator har ett speciellt andningsmönster med små variationer i andetagen. Därigenom varierar även den utandade mängden koldioxid marginellt över tid vilket används för att beräkna hur mycket hjärtat pumpar. Mätvärden från denna metod kommer att samlas in som ett komplement för att konstruera AI algoritmen. Metoden kommer också att utvärderas mot vår ordinarie metod för hjärt- och lungövervakning.

Vi kommer att ta blodprover, cirka 1-2 milliliter per gång, varje timme då operationen pågår för att analysera syremängden samt ett antal andra viktiga parametrar.

Det som beskrivs som skillnader ovan är inget som du märker av eller som påverkar dig, varken under operationen eller efteråt.

# Möjliga följder och risker med att delta i projektet

Det finns inga kända risker med det nya andningsmönstret, narkosmetoden, den speciellt anpassade ventilatorn eller extra provtagning under operation. Den har använts vid flera studier på människor tidigare. Det finns inga direkta fördelar förutom att din hjärtfunktion kommer att övervakas extra noga.

Du kan när som helst avbryta ditt deltagande i studien utan någon påverkan på vården i samband med din operation.

# Vad händer med mina uppgifter?

Projektet kommer att samla in och registrera information om dig. I samband med att du inkluderas i denna studie kommer vi inhämta grundläggande uppgifter om din sjukhistoria inklusive svar på aktuella laboratorieprover från sjukhusets journalsystem. Data från övervakningsutrustningen kommer att hämtas från sjukhuset krypterade lagring för patientövervakning och sparas i avidentifierad form. Vi studieansvariga som ansvarar för denna genomgång har tystnadsplikt. Uppgifterna om deltagande patienter kommer att kodas så att enskilda patienter inte kan identifieras av obehöriga. Uppgifter om deltagande patienter kommer att sparas av oss studieansvariga i enlighet med rutiner i upp till 10 år. Dina svar och resultat behandlas så att inte obehöriga kan ta del av dem. De avidentifierade resultaten av studien kommer sammanställas i syfte att publiceras i en medicinsk tidskrift, där vi endast kommer presentera avidentifierade data på gruppnivå.

Dina svar och dina resultat kommer att behandlas så att inte obehöriga kan ta del av dem.

Ansvarig för dina personuppgifter är Region Stockholm. Enligt EU:s dataskyddsförordning har du rätt att kostnadsfritt få ta del av de uppgifter om dig som hanteras i projektet, och vid behov få eventuella fel rättade. Du kan också begära att uppgifter om dig raderas samt att behandlingen av dina personuppgifter begränsas. Rätten till radering och till begränsning av behandling av personuppgifter gäller dock inte när uppgifterna är nödvändiga för den aktuella forskningen. Om du vill ta del av uppgifterna ska du kontakta Håkan Björne, Funktion PMI Karolinska Universitetssjukhuset Huddinge, telefon 08-123 800 00. Dataskyddsombud nås på e-mail: <a href="mailto:dataskyddsombud.karolinska@regionstockholm.se">dataskyddsombud.karolinska@regionstockholm.se</a>. Om du är missnöjd med hur dina personuppgifter behandlas har du rätt att ge in klagomål till Integritetsskyddsmyndigheten, som är tillsynsmyndighet.

#### Vad händer med mina prover?

Resultaten kommer att föras in i din journal.

## Hur får jag information om resultatet av projektet?

Om du är intresserad av att få reda på de data som lagrats om dig eller resultaten av hela studien är du välkommen att kontakta någon av oss ansvariga för studien. Du är välkommen att ta del av den vetenskapliga publikation som planeras.

# Försäkring och ersättning

För denna studie gäller patientförsäkringen. Ingen ersättning utgår.

# Deltagandet är frivilligt –anvisningar för att avbryta studien

Ditt deltagande är frivilligt och du kan när som helst välja att avbryta deltagandet. Om du väljer att inte delta eller vill avbryta ditt deltagande behöver du inte uppge varför, och det kommer inte heller att påverka din framtida vård eller behandling. Om du vill avbryta ditt deltagande ska du kontakta den ansvariga för projektet (se nedan). All data som samlats in från din medverkan i studien kommer då att raderas från vår databas.

## Ansvariga för projektet

Thorir Sigmundsson Funktion PMI

Karolinska Universitetssjukhuset Solna thorir.sigmundsson@regionstockholm.se

Tel: 08-123 700 00

Håkan Björne

Funktion PMI, B31

Karolinska Universitetssjukhuset Huddinge hakan.bjorne@regionstockholm.se

Tel: 08-585 800 00

Caroline Hällsjö Sander

Funktion PMI

Karolinska Universitetssjukhuset Solna Caroline.hallsjosander@regionstockholm.se

Tel: 08-123 700 00

Al hypotension study CIV-22-09-040666